CLINICAL TRIAL: NCT07050810
Title: Thera-Clean® Microbubbles System: A Pilot Study in Patients With Skin Diseases
Brief Title: Thera-Clean® Microbubbles System in Patients With Skin Diseases
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Amy Paller, Principal Investigator, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00223929
Record Dates: First submitted 2025-06-16; First posted 2025-07-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Epidermolysis Bullosa; Ichthyosis; Atopic Dermatitis; Psoriasis
MeSH Terms: conditions — Epidermolysis Bullosa; Ichthyosis; Dermatitis, Atopic; Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- At Home Bath with TheraClean device (Experimental): Participants treated with Thera-Clean Microbubbles bath system
  Interventions: Device: TheraClean

INTERVENTIONS:
Device: TheraClean — Begins after Week 0 visit and continues through Week 8. Participants will take at least 3 baths/week (20-30 minutes each bath) but may bathe daily, if desired.
  Other Names: Thera-Clean® Microbubbles bath system

SUMMARY:
Thera-Clean® Microbubble has proved to improve skin conditions in animals, however little research has been done regarding human subjects. Microbubble technology is a chemical-free therapeutic aimed at clearing foreign and organic matter from hair follicles, eliminating odors, and reducing itch. This hydrotherapy is said to aid in the healing process of inflamed and distressed tissue, relieve pain, and serve to remove contaminated tissue. This study will evaluate the change in skin conditions from the use of Thera-Clean® Microbubble for cleansing and debriding wounds from selected subjects focused on patients with inflammatory skin disease (epidermolysis bullosa, ichthyosis, atopic dermatitis and/or psoriasis). Proper wound care to prevent infection is vitally important for these patients and the options of therapeutics are limited. This study will evaluate the change in skin conditions from the use of Thera-Clean® Microbubble for cleansing and debriding lesional skin.

ELIGIBILITY:
Inclusion Criteria:

* Patients 2 years of age or above with psoriasis, atopic dermatitis/eczema, epidermolysis bullosa, or ichthyosis
* Skin conditions to be stable for at least the previous 4-week period (patients will continue to use their typical skin treatment regimen throughout the study)

Exclusion Criteria:

* Patients with unstable skin conditions
* Patients not willing to comply with the study requirements for bathing at home
* Patients younger than 2 years of age

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Improvement of skin condition between baseline to Week 4 and baseline to Week 8 using Thera-Clean® microbubble bathing therapy as assessed by the Investigator Global Assessment (IGA). | 8 weeks
  IGA will be assessed on a 4-point scale: clear; almost clear; mild; moderate; severe.

SECONDARY OUTCOMES:
Change in subject's/proxy's perceived visibility and severity of skin disease as assessed by subject reported severity and visibility questionnaires. | 8 weeks
  assessed between baseline and Week 4 and Week 8
Overall improvement in the Dermatology Life Quality Index (>16 yo)/ Children or Proxy-reported Children Dermatology Life Quality Index (4-15 yo)/ Proxy-reported Infant Dermatology Life Quality Index (CDLQI/DLQI/IDLQI) (<4 yo) | 8 weeks
  assessed between baseline and Week 4 and Week 8
Change in Peak Pruritus/Pain Numeric Rating Scale and Peak Pain Numeric Rating Scale scores (0-10 scale) | 8 weeks
  assessed between baseline and Week 4 and Week 8
Change in odor as assessed by subject reported odor assessment questionnaires. | 8 weeks
  assessed between baseline and Week 4 and Week 8
Overall tolerability of device / device usage throughout study as assessed by subject reported tolerability survey. | 8 weeks
  assessed throughout the study
Overall satisfaction of device / device usage as assessed by subject reported satisfaction survey. | 8 weeks
  assessed throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Amy Paller, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Department of Dermatology, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No